CLINICAL TRIAL: NCT05210582
Title: An Open Label, Phase II Study to Assess the Changes in Pigmentation and Safety of Subcutaneous, Bioresorbable Afamelanotide Implants in the Treatment of Vitiligo on the Face
Brief Title: A Study to Assess the Changes in Pigmentation and Safety of Afamelanotide in Patients With Vitiligo on the Face
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinuvel, Inc. (Industry)
Responsible Party: Sponsor
Organization: Clinuvel Pharmaceuticals Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUV104
Record Dates: First submitted 2022-01-11; First posted 2022-01-27 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — afamelanotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Afamelanotide (Experimental)
  Interventions: Drug: Afamelanotide

INTERVENTIONS:
Drug: Afamelanotide — Patients will receive afamelanotide over a three-month period, with an additional three-month follow up.

SUMMARY:
The CUV104 study will assess the efficacy and safety of afamelanotide in patients with vitiligo on the face and body as a monotherapy in repigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a confirmed diagnosis of vitiligo on the face and with T-VASI range 0.5-50%
* Stable face vitiligo with F-VASI of at least 0.1%
* Stable or slowly progressive vitiligo over a 3-month period
* Fitzpatrick skin types IV-VI
* Treatment with narrowband (NB)-UVB light 2-3 times per week during the last four weeks preceding the first implant for priming

Exclusion Criteria:

* Patients with segmental vitiligo
* Fitzpatrick skin types I-III
* Treatment with NB-UVB phototherapy in the last three months prior to phototherapy, excluding the sessions for priming in the four weeks prior to treatment. A 3-month washout period from phototherapy is necessary prior to priming.
* Previous topical treatment for vitiligo
* Allergy to afamelanotide or the polymer contained in the implant or to lignocaine/lidocaine or other local anaesthetic to be used during the administration of the implant
* History of melanoma or lentigo maligna
* Any current skin disease that may interfere with the study evaluation
* Presence of severe hepatic disease or hepatic impairment
* Renal impairment
* History of systemic or psychiatric disease judged to be clinically significant by the Investigator and which may interfere with the study evaluation
* Female who is pregnant or lactating
* Female of child-bearing potential not using adequate contraceptive measures during the treatment phase and for a period of three months thereafter
* Sexually active man with a partner of child-bearing potential who is not using adequate contraceptive measures, as described above
* Participation in a clinical trial for an investigational agent within 30 days prior to the Screening Visit
* Use of any other prior and concomitant therapy which may interfere with the objective of the study
* Subjects assessed as not suitable for the study in the opinion of the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving Vitiligo Area Scoring Index (VASI)25 on facial lesions | From Baseline to Day 84
  Measured using Vitiligo Area Scoring Index (VASI). A decrease in VASI indicates a reduction of the facial surface area affected by vitiligo (possible range 1-100)

SECONDARY OUTCOMES:
Proportion of participants achieving Vitiligo Area Scoring Index (VASI)25 on body surface area | From Baseline to Day 84
  Proportion of participants achieving VASI25 on body surface area (excluding hands and feet). A decrease in VASI indicates a reduction of the facial surface area affected by vitiligo (possible range 1-100).
Percentage change in pigmentation on body surface area measured by the VASI scoring system | From Baseline to Day 84
  Percentage change in pigmentation on body surface area (excluding hands and feet) measured by VASI scoring system. A decrease in VASI indicates a reduction of the body surface area affected by vitiligo (possible range 1-100)
Percentage change in pigmentation on facial surface area measured by the VASI scoring system | From Baseline to Day 168
  A decreased VASI indicates a reduction in the faces' degree of depigmentation (possible range 1-100)
Change in Perception of Vitiligo Severity using a vitiligo validated specific tool (A) | From Baseline to Day 168
  The higher the score, the more severe the disease
Change in Noticeability of Vitiligo using a vitiligo validated specific tool (B) | From Baseline to Day 168
  Higher the value means lower noticeability
Change in Quality of life using a vitiligo specific tool (C) | From Baseline to Day 168
  Higher value means a lower quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- CLINUVEL Investigational site, Detroit, Michigan, United States